CLINICAL TRIAL: NCT04982822
Title: Novel Senhance Robotic System in Urologic Surgery: Its Clinical Application and Implication
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202004072RINA
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Urologic Diseases; Surgery
Keywords: Urology; Senhance; Robotic surgical system; Laparoscopic surgery
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An observational study to collect data from the participants who received urologic surgeries using the Senhance Robotic system.

DETAILED DESCRIPTION:
This is an observational study and investigators will collect peri-operative demographic data, and short-term outcomes (3-6 months) from the participants who received minimal invasive surgeries using Senhance robotic system in the National Taiwan University Hospital Yunlin Branch, Urology Department. The investigators want to demonstrate if the robotic system is safe and feasible in urologic laparoscopic surgeries.

The operation included TEP, radical prostatectomy, radical nephrectomy (nephroureterectomy) , adrenalectomy, radical cystectomy, and ureter surgery et al.

up to 2022/12, we had recruited 127 TEP, 83 radical prostatectomies, 17 adrenalectomies, 40 nephrectomies, 29 partial nephrectomies, 13 radical cystectomies and 18 other surgeries, such as ureter surgery

ELIGIBILITY:
Patients undergo laparoscopic urologic surgeries

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study populations consisted of aged from 18 years old to 90 years old and had will to receive laparoscopic surgeries using the Senhance robotic system.
  The were excluded if there's major severe cardio-pulmonary condition or had received extensive abdominal surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Peri-operative complications | postoperative 30 days
  Using Clavien-Dindo classification to record the safety outcome
short-term outcome | 3-6 months
  the short-term outcome was according to a different surgery, such as post-operative 3 months PSA, incontinence rate in radical prostatectomy,

CONTACTS AND LOCATIONS:
Overall Officials: LunHsiang Yuan, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Outside U.S./Canada, Taiwan